CLINICAL TRIAL: NCT02466087
Title: Role of Magnesium Supplementation in the Treatment of Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Emily Tarleton, Bionutrition Research Manager, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M15-337
Record Dates: First submitted 2015-05-29; First posted 2015-06-09 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mg Cl (Experimental): 500mg Mg Cl per day for 6 weeks
  Interventions: Drug: Mg Cl
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Mg Cl — Four supplements a day for 6 weeks.
  Arms: Mg Cl

SUMMARY:
The objective of this project is to test the hypothesis that magnesium supplementation will decrease depressive symptoms in adults.

This study takes place over 12 consecutive weeks. While the investigators will follow the volunteers for the full 12 weeks volunteers will only take magnesium supplements for 6 consecutive weeks. Volunteers will be randomly assigned to start the supplement at week 1 or week 7. Volunteers will take two supplement two times a day for a total of 248 mg elemental magnesium daily in the form of magnesium chloride. This amount of magnesium is less than the tolerable upper limit of 350 mg per day. The supplements will be provided. Volunteers will be asked to maintain their normal diet for the 12 weeks of the study.

The primary outcome measure is the PHQ-9 questionnaire, a validated measure of depression. Secondary measures include the GAD-7 for Anxiety and side effects.

ELIGIBILITY:
Inclusion Criteria:

* All adults at least 18 years of age
* A Patient Health Questionnaire-9 (PHQ-9) score of greater or equal to 5 but less than 20
* People who are currently being treated for depression are still eligible to participate but their treatment must be stable (no changes in medication dose or brand and/or no changes in therapy regimen for at least 2 months).

Exclusion Criteria:

* Active delirium or dementia
* Medicinal treatment for bipolar disorder, personality disorder or schizophrenia,
* Glomerular Filtration Rate of less than 60
* Irritable Bowel Disease
* Inflammatory Bowel Disease
* GERD
* Gastritis
* Pregnant as reported by potential volunteer
* Myasthenia Gravis
* Planned elective surgery
* Currently taking

  * Long Term Antibiotics
  * Fluoroquinolone
  * Trientine or Penicillamine
  * Long Term Antivirals
  * Digoxin
  * Bisphosphonates
  * Eltrombopag
  * Opiods
  * Calcium Channel Blockers
  * Deferiprone
  * Doxercalciferol
* Unable or unwilling to stop taking a magnesium supplement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Tarleton, MS, RD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mg Cl (Weeks 1-6), Then no Intervention (Weeks 7-12): MgCl for weeks 1-6 and then no treatment for weeks 7-12
- No Intervention (Weeks 1-6), Then MgCl (Weeks 7-12): No Treatment for weeks 1-6 and then MgCl for weeks 7-12
Period: First Intervention: Weeks 1-6
Arm/Group | Mg Cl (Weeks 1-6), Then no Intervention (Weeks 7-12) | No Intervention (Weeks 1-6), Then MgCl (Weeks 7-12)
Started | 62 | 64
Completed | 55 | 57
Not Completed | 7 | 7
Period: Second Intervention: Weeks 7-12
Arm/Group | Mg Cl (Weeks 1-6), Then no Intervention (Weeks 7-12) | No Intervention (Weeks 1-6), Then MgCl (Weeks 7-12)
Started | 55 | 57
Completed | 55 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive MgCl first and no intervention first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 126
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Numbers represent participants with analyzable data.
  years | 52.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Numbers reflect participants with analyzable data
  Participants
    Female | 78
    Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 123
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 126

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire-9
Description: Change in score from week 1 to week 6 and week 7 to week 12 (difference in differences)
  The Patient Health Questionnaire-9 Item is a validated questionnaire with high sensitivity and specificity for the diagnosis of depression. The PHQ-9 score can range from 0 to 27, with the following severity scores: 0-4 None; 5-9 Mild; 10-14 Moderate; 15-19 Moderate to Severe; 20-27 Severe.
Time Frame: 12 weeks
Population: Number of participants with analyzable data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- MgCl: 6 weeks of MgCl supplements
- Control: 6 weeks of no supplements
Arm/Group | MgCl | Control
Number analyzed (Participants) | 112 | 112
score on a scale | -4.28 [-4.99 to -3.56] | -0.09 [-0.90 to 0.72]
Statistical Analysis 1: Comparison: MgCl vs Control; Test type: Other; Regression, Linear; diiference in differences = 1.5

2. Secondary Outcome: Generalized Anxiety Disorder 7 Item Questionnaire
Description: Change in score from week 1 to week 6 and week 7 to 12 (difference in differences)
  GAD-7 score has been shown to be a valid indication of anxiety symptoms. The GAD-7 score can range from 0 to 21, with the following severity scores: 0-4 None; 5-9 Mild; 10-14 Moderate; 15-21 Severe.
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Groups:
- MgCl: 6 weeks of MgCl supplementation
Arm/Group | MgCl | Control
Number analyzed (Participants) | 112 | 112
scores on a scale | -3.88 [-4.70 to -3.07] | 0.80 [0.02 to 1.59]

3. Secondary Outcome: Change in Headaches While Taking Supplements
Description: Change in headaches compared to normal during the 6 weeks on supplements. Change was calculated from 2 time points-start of supplements and end of supplements.
  Change was recorded as 0, None (same)
  1. Mild
  2. Moderate
  3. Severe (worse)
Time Frame: 12 weeks
Population: headaches
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MgCl | Control
Number analyzed (Participants) | 112 | 112
score on a scale | -0.14 [-0.25 to -0.03] | -0.14 [-0.25 to -0.03]

ADVERSE EVENTS:
Groups:
- Mg Supplementation: 6 weeks of Mg Supplements
- Control: 6 weeks of no MgCl supplements
Arm/Group | Mg Supplementation | Control
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/64
Other Adverse Events (participants affected / at risk) | 0/62 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-04-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT02466087/Prot_000.pdf
  • Informed Consent Form (2016-01-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT02466087/ICF_001.pdf